CLINICAL TRIAL: NCT00279201
Title: The Durability of Twice-Daily Insulin Lispro Low Mixture Compared to Once-Daily Insulin Glargine When Added to Existing Oral Therapy in Patients With Type 2 Diabetes and Inadequate Glycemic Control
Brief Title: The DURABLE Trial: Evaluating the Durability of Starter Insulin Regimens in Patients With Type 2 Diabetes (IOOV)
Acronym: IOOV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10455; F3Z-US-IOOV (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-12-15; First posted 2006-01-19 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin Glargine; insulin lispro, isophane insulin lispro drug combination (25:75); Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Insulin glargine (Active Comparator): Initiation Phase: Insulin glargine for 24 weeks Maintenance: Up to an additional 2 years of insulin glargine if glycosylated hemoglobin (HbA1c) less than or equal to 7.0 at 24 weeks.
  Interventions: Drug: Insulin glargine
- Lispro Low Mix (Experimental): Initiation Phase: Lispro Low Mix (LM) for 24 weeks Maintenance Phase: Up to an additional 2 years of Lispro LM if HbA1c less than or equal to 7.0 at 24 weeks.
  Interventions: Drug: Lispro Low Mix
- Lispro Mid Mix prior Lispro Low Mix addendum (Experimental): Following Lispro LM Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, participants could be randomized to receive Lispro Mid Mix for 24 weeks in the Intensification Addendum Phase.
  Interventions: Drug: Lispro Mid Mix
- Lispro Low Mix prior Glargine addendum (Experimental): Following Insulin Glargine Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, participants could be randomized to receive Lispro Low Mix for 24 weeks in the Intensification Addendum Phase
  Interventions: Drug: Lispro Low Mix
- Basal bolus prior Lispro Low Mix addendum (Active Comparator): Following Lispro LM Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, participants could be randomized to receive Basal Bolus therapy (combination of insulin glargine and lispro) for 24 weeks in the Intensification Addendum Phase.
  Interventions: Drug: Insulin glargine; Drug: Lispro
- Basal bolus prior Glargine addendum (Active Comparator): Following Insulin Glargine Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, participants could be randomized to receive Basal Bolus therapy (combination of insulin glargine and lispro) for 24 weeks in the Intensification Addendum Phase.
  Interventions: Drug: Insulin glargine; Drug: Lispro

INTERVENTIONS:
Drug: Insulin glargine — Subcutaneous injection daily
  Other Names: Lantus
  Arms: Basal bolus prior Glargine addendum; Basal bolus prior Lispro Low Mix addendum; Insulin glargine
Drug: Lispro Low Mix — Subcutaneous injection twice daily.
  Other Names: Humalog Mix 75/25
  Arms: Lispro Low Mix; Lispro Low Mix prior Glargine addendum
Drug: Lispro Mid Mix — Lispro Mid Mix subcutaneous injection 3 times daily.
  Other Names: Humalog Mix 50/50
  Arms: Lispro Mid Mix prior Lispro Low Mix addendum
Drug: Lispro — Lispro subcutaneous injection 3 times daily.
  Other Names: Humalog
  Arms: Basal bolus prior Glargine addendum; Basal bolus prior Lispro Low Mix addendum

SUMMARY:
This study will compare insulin lispro low mixture [LM] and insulin glargine both in combination with the patient's oral diabetes medicines, for their ability to control blood sugar in patients with type 2 diabetes and compare insulin lispro LM to insulin glargine with regard to the length of time that the overall blood sugar can be controlled.

This study will also determine whether the safety of insulin lispro LM and any side effects that might be associated with it are different from those observed with insulin glargine, both in combination with the patient's oral diabetes medications.

The addendum study (Intensification Addendum) will compare how different insulin treatments work to control blood sugar in patients whose diabetes could not be controlled by either insulin lispro LM or insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* Must have type 2 diabetes.
* Must be at least 30 and less than 80 years of age at the time of Visit 1.
* Must be on at least two oral antidiabetes medications for at least 90 days.
* Must have an HbA1c 1.2 to 2.0 times the upper limit of normal reference range at the local lab.

Exclusion Criteria:

* Must not have used insulin on a regular basis in the last 12 months.
* Must not have had more than one episode of severe hypoglycemia in the last 24 weeks.
* Must not have a body mass index (BMI) of greater than 45 (morbid obesity).
* Must not have clinically significant hematologic, oncologic, renal, cardiac, hepatic, or gastrointestinal disease.
* Must not be pregnant or intend to get pregnant during course of the study.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2091 (Actual)
Dates: Start 2005-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (199):
- United States (138):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mobile, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Litchfield Park, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlingame, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fountain Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Jolla, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Mesa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Alamitos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Gatos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwalk, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salinas, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vacaville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ventura, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cromwell, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Deerfield Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Inverness, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kissimmee, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Worth, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Melbourne, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winter Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kellogg, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belleville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gurnee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., O'Fallon, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Wayne, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bowling Green, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madisonville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Owensboro, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elkridge, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elkton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reisterstown, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Towson, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Haverhill, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waltham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomfield Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Troy, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesterfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cherry Hill, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flemington, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stratford, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teaneck, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cooperstown, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mamaroneck, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Massapequa, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hartford, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westfield, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Huntersville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morganton, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tabor City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jamestown, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akron, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Franklin, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medford, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fleetwood, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Levittown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hartsville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnson City, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingsport, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Abilene, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Paso, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Killeen, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midland, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Braunfels, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogden, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Provo, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellingham, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Everett, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Renton, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wenatchee, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eau Claire, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marshfield, Wisconsin
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mar del Plata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pilar
- Australia (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingswood Penrith, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Keswick, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burnie, Tasmania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nedlands, Western Australia
- Brazil (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Curitiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., SÃ£o Paulo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Setor Oeste/Goiania
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Red Deer, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Petitcodiac, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ajax, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mississauga, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niagara Falls, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Laval, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Greece (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nikaias - Piraeus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eger
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szekszárd
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szentes
- India (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ahemdabad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aligarh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coimbatore
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyderabaad
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Karnal/Haryana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trivandrum
- Netherlands (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brunssum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Emmen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoogeveen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Venlo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwijndrecht
- Puerto Rico (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orcorvis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- Romania (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Târgu Mureş
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dos Hermanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mosteles
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Requena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander

REFERENCES:
- [Result] Herman WH, Dungan KM, Wolffenbuttel BH, Buse JB, Fahrbach JL, Jiang H, Martin S. Racial and ethnic differences in mean plasma glucose, hemoglobin A1c, and 1,5-anhydroglucitol in over 2000 patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 May;94(5):1689-94. doi: 10.1210/jc.2008-1940. Epub 2009 Mar 10. PMID 19276235
- [Result] Fahrbach J, Jacober S, Jiang H, Martin S. The DURABLE trial study design: comparing the safety, efficacy, and durability of insulin glargine to insulin lispro mix 75/25 added to oral antihyperglycemic agents in patients with type 2 diabetes. J Diabetes Sci Technol. 2008 Sep;2(5):831-8. doi: 10.1177/193229680800200514. PMID 19885269
- [Derived] Scheen AJ, Schmitt H, Jiang HH, Ivanyi T. Individualizing treatment of type 2 diabetes by targeting postprandial or fasting hyperglycaemia: Response to a basal vs a premixed insulin regimen by HbA1c quartiles and ethnicity. Diabetes Metab. 2015 Jun;41(3):216-22. doi: 10.1016/j.diabet.2015.03.002. Epub 2015 Apr 14. PMID 25881510
- [Derived] Jovanovic L, Peters AL, Jiang HH, Hardin DS. Durability of glycemic control with insulin lispro mix 75/25 versus insulin glargine for older patients with type 2 diabetes. Aging Clin Exp Res. 2014 Apr;26(2):115-21. doi: 10.1007/s40520-013-0140-8. Epub 2013 Oct 3. PMID 24092662
- [Derived] Wolffenbuttel BH, Herman WH, Gross JL, Dharmalingam M, Jiang HH, Hardin DS. Ethnic differences in glycemic markers in patients with type 2 diabetes. Diabetes Care. 2013 Oct;36(10):2931-6. doi: 10.2337/dc12-2711. Epub 2013 Jun 11. PMID 23757434
- [Derived] Qu Y, Jacober SJ, Zhang Q, Wolka LL, DeVries JH. Rate of hypoglycemia in insulin-treated patients with type 2 diabetes can be predicted from glycemic variability data. Diabetes Technol Ther. 2012 Nov;14(11):1008-12. doi: 10.1089/dia.2012.0099. PMID 23101951
- [Derived] Buse JB, Wolffenbuttel BH, Herman WH, Hippler S, Martin SA, Jiang HH, Shenouda SK, Fahrbach JL. The DURAbility of Basal versus Lispro mix 75/25 insulin Efficacy (DURABLE) trial: comparing the durability of lispro mix 75/25 and glargine. Diabetes Care. 2011 Feb;34(2):249-55. doi: 10.2337/dc10-1701. PMID 21270182
- [Derived] Miser WF, Arakaki R, Jiang H, Scism-Bacon J, Anderson PW, Fahrbach JL. Randomized, open-label, parallel-group evaluations of basal-bolus therapy versus insulin lispro premixed therapy in patients with type 2 diabetes mellitus failing to achieve control with starter insulin treatment and continuing oral antihyperglycemic drugs: a noninferiority intensification substudy of the DURABLE trial. Clin Ther. 2010 May;32(5):896-908. doi: 10.1016/j.clinthera.2010.05.001. PMID 20685497
- [Derived] Wolffenbuttel BH, Klaff LJ, Bhushan R, Fahrbach JL, Jiang H, Martin S. Initiating insulin therapy in elderly patients with Type 2 diabetes: efficacy and safety of lispro mix 25 vs. basal insulin combined with oral glucose-lowering agents. Diabet Med. 2009 Nov;26(11):1147-55. doi: 10.1111/j.1464-5491.2009.02824.x. PMID 19929994
- [Derived] Buse JB, Wolffenbuttel BH, Herman WH, Shemonsky NK, Jiang HH, Fahrbach JL, Scism-Bacon JL, Martin SA. DURAbility of basal versus lispro mix 75/25 insulin efficacy (DURABLE) trial 24-week results: safety and efficacy of insulin lispro mix 75/25 versus insulin glargine added to oral antihyperglycemic drugs in patients with type 2 diabetes. Diabetes Care. 2009 Jun;32(6):1007-13. doi: 10.2337/dc08-2117. Epub 2009 Mar 31. PMID 19336625
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Initiation: Glargine or Lispro LM - 24 weeks. Maintenance: Up to 2 more years treatment if HbA1c <=7.0 at 24 weeks. After Initiation, if HbA1c >7.0 after 24 weeks, instead of entering Maintenance, those from Lispro LM could receive Basal bolus or Mid Mix; glargine could receive Basal bolus or Lispro LM for 24 weeks in Intensification Addendum.
Groups:
- Insulin Glargine: Initiation Phase: Insulin glargine for 24 weeks. Maintenance: Up to an additional 2 years of insulin glargine if glycosylated hemoglobin (HbA1c) less than or equal to 7.0 at 24 weeks.
- Lispro Low Mix: Initiation Phase: Lispro Low Mix (LM) for 24 weeks. Maintenance Phase: Up to an additional 2 years of Lispro LM if HbA1c less than or equal to 7.0 at 24 weeks.
- Lispro Mid Mix Prior Lispro Low Mix Addendum: Following Lispro LM Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, they could be randomized to receive Lispro Mid Mix for 24 weeks in the Intensification Addendum Phase.
- Lispro Low Mix Prior Glargine Addendum: Following Insulin Glargine Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, they could be randomized to receive Lispro Low Mix for 24 weeks in the Intensification Addendum Phase.
- Basal Bolus Prior Lispro Low Mix Addendum: Following Lispro LM Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, they could be randomized to receive Basal Bolus therapy (combination of insulin glargine and lispro) for 24 weeks in the Intensification Addendum Phase.
- Basal Bolus Prior Glargine Addendum: Following Insulin Glargine Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, they could be randomized to receive Basal Bolus therapy (combination of insulin glargine and lispro) for 24 weeks in the Intensification Addendum Phase.
Period: Initiation
Arm/Group | Insulin Glargine | Lispro Low Mix | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro Low Mix Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Started | 1046 | 1045 | 0 | 0 | 0 | 0
Completed | 918 | 900 | 0 | 0 | 0 | 0
Not Completed | 128 | 145 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 5 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 15 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 42 | 41 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Exclusion | 7 | 9 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 9 | 10 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 35 | 41 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 15 | 18 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 13 | 5 | 0 | 0 | 0 | 0
Not completed — Discontinuation Oral Antihyperglycemics | 0 | 1 | 0 | 0 | 0 | 0
Period: Maintenance
Arm/Group | Insulin Glargine | Lispro Low Mix | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro Low Mix Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Started | 419 (100 left the study after initiation. 399 had HbA1c>7% and enrolled in intensification addendum.) | 473 (82 left the study after initiation. 345 had HbA1c>7% and enrolled in intensification addendum.) | 0 | 0 | 0 | 0
Completed | 188 | 239 | 0 | 0 | 0 | 0
Not Completed | 231 | 234 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 32 | 30 | 0 | 0 | 0 | 0
Not completed — Discontinuation Antihyperglycemic Drugs | 3 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Death | 4 | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 17 | 13 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Exclusion | 1 | 4 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 16 | 24 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 18 | 18 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 9 | 9 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 4 | 0 | 0 | 0 | 0 | 0
Not completed — HbA1c>7.5% | 123 | 126 | 0 | 0 | 0 | 0
Period: Intensification Addendum
Arm/Group | Insulin Glargine | Lispro Low Mix | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro Low Mix Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Started | 0 | 0 | 174 | 200 | 171 | 199
Completed | 0 | 0 | 151 | 172 | 142 | 162
Not Completed | 0 | 0 | 23 | 28 | 29 | 37
Not completed — Withdrawal by Subject | 0 | 0 | 12 | 14 | 9 | 18
Not completed — Lost to Follow-up | 0 | 0 | 4 | 6 | 7 | 7
Not completed — Protocol Violation | 0 | 0 | 2 | 2 | 6 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 4 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 4 | 1 | 3 | 2
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Entry Criteria Exclusion | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lispro LM: Initiation Phase: Lispro Low Mix (LM) for 24 weeks. Maintenance Phase: Up to an additional 2 years of Lispro LM if HbA1c less than or equal to 7.0 at 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine | Lispro LM | Total
Number analyzed (Participants) | 1046 | 1045 | 2091
Age Continuous [Mean (Standard Deviation); unit: years] | 56.59 (9.95) | 57.05 (9.73) | 56.82 (9.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 493 | 987
  Male | 552 | 552 | 1104
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 668 | 651 | 1319
  African Descent | 70 | 62 | 132
  East/Southeast Asian | 27 | 18 | 45
  Hispanic | 116 | 136 | 252
  Other | 29 | 39 | 68
  Western Asian | 136 | 139 | 275
Region of Enrollment [Number; unit: participants]
  United States | 509 | 513 | 1022
  Hungary | 24 | 26 | 50
  Greece | 25 | 25 | 50
  Canada | 60 | 60 | 120
  Argentina | 98 | 95 | 193
  Brazil | 45 | 46 | 91
  Spain | 47 | 49 | 96
  Romania | 29 | 28 | 57
  Australia | 48 | 48 | 96
  Netherlands | 30 | 27 | 57
  India | 131 | 128 | 259
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 88.23 (20.78) | 88.84 (20.97) | 88.53 (20.87)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meters squared (kg/m^2)] | 31.69 (6.01) | 31.67 (5.96) | 31.68 (5.98)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 9.30 (5.93) | 9.73 (6.29) | 9.51 (6.11)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent glycosylated hemoglobin] | 9.02 (1.24) | 9.06 (1.29) | 9.04 (1.26)
1,5 Anhydroglucitol (1,5 AG) [Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)] | 4.97 (4.06) | 5.02 (4.12) | 4.99 (4.09)
Mean of Pre-Meals Blood Glucose [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 201.29 (57.40) | 198.97 (54.87) | 200.13 (56.14)
Mean of Post Meals Blood Glucose (Postprandial) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 241.58 (61.06) | 240.08 (58.15) | 240.82 (59.61)
Average of All Blood Glucose [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 218.05 (56.55) | 216.12 (54.40) | 217.08 (55.48)
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 196.16 (55.14) | 192.91 (53.22) | 194.53 (54.20)

OUTCOME MEASURES:

1. Primary Outcome: INITIATION: 24-Week Endpoint Glycosylated Hemoglobin (HbA1c)
Time Frame: Endpoint (Initiation: Week 24)
Population: Last observation carried forward (LOCF) method was performed on the intent-to-treat (ITT) population who had at least 1 post-baseline assessment in the initiation phase. Initiation baseline: Week 0.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Groups:
- Insulin Glargine: Insulin glargine for 24 weeks.
- Lispro Low Mix: Lispro Low Mix (LM) for 24 weeks.
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 990 | 986
percent glycosylated hemoglobin | 7.33 (1.07) | 7.23 (1.08)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.005, ANCOVA; P-value from ANCOVA, baseline value as covariate. Response = Treatment + Baseline + Country + thiazolidinedione (TZD) use + Sulfonylurea (sulfo) use

2. Primary Outcome: MAINTENANCE: Duration of Time HbA1c Maintained at Goal by Initiation Regimen (Insulin Glargine or Lispro Low Mix)
Description: HbA1c goal: HbA1c ≤7.0% or HbA1c >7.0% but increased <0.4% from last HbA1c ≤7.0%
Time Frame: Endpoint (Last Observation Carried Forward [LOCF]) (Maintenance: up to 2.5 years)
Population: Last observation carried forward method was performed on the intent-to-treat (ITT) population who had at least 1 post-baseline assessment. Maintenance baseline: Week 24.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Insulin Glargine: Maintenance Phase: Up to an additional 2 years of insulin glargine if glycosylated hemoglobin (HbA1c) less than or equal to 7.0 at 24 weeks.
- Lispro Low Mix: Maintenance Phase: Up to an additional 2 years of Lispro LM if HbA1c less than or equal to 7.0 at 24 weeks.
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 418 | 470
months | 14.40 [13.40 to 16.83] | 16.80 [14.03 to 19.67]
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.040, Log Rank; Stratified by country, thiazolidinedione (TZD) use, sulfo use

3. Primary Outcome: ADDENDUM: 24-Week Endpoint HbA1c
Description: HbA1c at 24-week endpoint in Intensification Addendum of the trial.
Time Frame: Endpoint (Addendum) (24 weeks: Week 48)
Population: Last observation carried forward (LOCF) method was performed on the intent-to-treat (ITT) population who had at least 1 post-baseline assessment. Addendum baseline: Week 24: 48 weeks.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Groups:
- Lispro LM Prior Glargine Addendum: Following Insulin Glargine Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, they could be randomized to receive Lispro Low Mix for 24 weeks in the Intensification Addendum Phase.
Arm/Group | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro LM Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Number analyzed (Participants) | 160 | 187 | 159 | 176
percent glycosylated hemoglobin | 8.19 (1.26) | 8.03 (1.15) | 8.16 (1.43) | 8.14 (1.53)
Statistical Analysis 1: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.271, ANCOVA; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 2: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.990, ANCOVA; Response = Treatment + Baseline + Country + TZD use

4. Secondary Outcome: INITIATION: Change in HbA1c From Baseline to 24 Weeks
Time Frame: Baseline (Initiation) to Endpoint (LOCF, Week 24)
Population: Last observation carried forward (LOCF) method was performed on the intent-to-treat (ITT) population who had at least 1 post-baseline assessment. Initiation baseline: Week 0.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 977 | 962
percent glycosylated hemoglobin | -1.68 (1.27) | -1.83 (1.27)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.005, ANCOVA; Response = Treatment + Baseline + Country + TZD use + Sulfo use

5. Secondary Outcome: INITIATION: Percentage of Participants With HbA1c < or = 7.0%, HbA1c <7.0%, and HbA1c < or = 6.5% at Endpoint
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 990 | 986
percentage of participants
  <=7.0% | 45.8 | 52.5
  <7.0% | 40.3 | 47.5
  <=6.5% | 22.2 | 24.6
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — P-value for <=7.0%; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is for <7.0%; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.174, Cochran-Mantel-Haenszel — P-value is for <=6.5%; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use

6. Secondary Outcome: INITIATION: HbA1c
Time Frame: Baseline (Initiation), Week 12, Week 24, Endpoint (LOCF)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 1030 | 1017
percent glycosylated hemoglobin
  Baseline (n=1030,1017) | 9.02 (1.24) | 9.06 (1.29)
  Week 12 (n=952,953) | 7.42 (0.95) | 7.27 (0.99)
  Week 24 (n=922,911) | 7.28 (1.06) | 7.19 (1.03)
  Endpoint (LOCF) (n=990,986) | 7.33 (1.07) | 7.23 (1.08)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.416, ANOVA — P-value for baseline; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Week 12; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value for Week 24; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value for endpoint; Response = Treatment + Baseline + Country + TZD use + sulfo use

7. Secondary Outcome: INITIATION: 7-point Self-monitored Plasma Glucose (SMPG) Profiles and Postprandial Excursions
Description: Abbreviations: AM = morning; BG = blood glucose; PM = evening; PP = postprandial. A postprandial excursion is defined as: 2 hour postmeal plasma glucose-premeal plasma glucose.
Time Frame: Endpoint (LOCF) (Initiation: Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams per 100 Milliliters (mg/dL)
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 989 | 995
milligrams per 100 Milliliters (mg/dL)
  Baseline mean fasting blood glucose (n=986,993) | 196.16 (55.14) | 192.91 (53.22)
  Mean fasting blood glucose (n=938,922) | 121.52 (33.41) | 133.54 (35.00)
  Baseline AM 2-hour postprandial BG (n=977,989) | 251.45 (64.78) | 252.46 (64.54)
  AM 2-hour postprandial blood glucose (n=932,920) | 171.79 (49.14) | 167.40 (49.46)
  Baseline midday premeal BG (n=976,988) | 203.87 (67.31) | 203.76 (65.93)
  Midday premeal blood glucose (BG) (n=934,919) | 137.43 (44.05) | 130.36 (42.44)
  Baseline midday 2-hour postprandial BG (n=974,988) | 232.73 (68.84) | 231.53 (66.18)
  Midday 2-hour postprandial BG (n=929,916) | 169.38 (46.78) | 167.91 (48.00)
  Baseline evening pre-meal BG (n=983,993) | 203.33 (66.50) | 200.36 (64.56)
  Evening pre-meal blood glucose (n=936,922) | 141.86 (45.44) | 143.44 (43.09)
  Baseline evening 2hour postprandial BG (n=983,991) | 239.73 (70.28) | 236.33 (64.92)
  Evening 2-hour postprandial BG (n=932,921) | 175.73 (48.66) | 163.20 (46.67)
  Baseline 3 AM blood glucose (n=955,975) | 197.99 (64.28) | 194.11 (61.96)
  3 AM blood glucose (n=912,899) | 131.08 (42.38) | 129.70 (40.51)
  Baseline AM 2-hour BG excursion (n=975,987) | 55.32 (46.93) | 60.06 (47.21)
  AM 2-hour blood glucose excursion (n=932,920) | 50.57 (43.59) | 34.01 (45.04)
  Baseline midday 2-hour BG excursion (n=966,981) | 26.60 (48.50) | 28.08 (45.09)
  Midday 2-hour blood glucose excursion (n=928,916) | 32.21 (40.40) | 37.46 (44.40)
  Baseline PM 2-hour BG excursion (n=979,988) | 36.50 (46.11) | 36.31 (44.37)
  PM 2-hour blood glucose excursion (n=929,921) | 34.17 (40.30) | 19.51 (42.90)
  Baseline mean all meal time excursions (n=985,991) | 40.80 (29.92) | 41.63 (28.58)
  Mean of all meal time excursions (n=935,921) | 38.96 (27.22) | 30.34 (28.22)
  Baseline mean all 2hour PP BG (n=986,993) | 241.58 (61.06) | 240.08 (58.15)
  Mean of all 2-hour postprandial BG (n=935,921) | 172.28 (41.04) | 166.17 (39.82)
  Baseline AM/PM 2-hour postprandial BG (n=986,993) | 245.67 (62.02) | 244.36 (59.24)
  AM/PM 2-hour postprandial BG (n=935,921) | 173.73 (42.83) | 165.19 (41.71)
  Baseline mean all premeal BG (n=988,994) | 201.29 (57.40) | 198.97 (54.87)
  Mean of all premeal blood glucose (n=938,922) | 133.62 (34.09) | 135.80 (32.80)
  Baseline AM/PM 2-hour BG excursion (n=985,991) | 46.05 (35.06) | 48.11 (35.77)
  AM/PM 2-hour blood glucose excursion (n=935,921) | 42.42 (31.96) | 26.74 (34.01)
  Baseline mean of all BG values (n=989,995) | 218.05 (56.55) | 216.12 (54.40)
  Mean of all blood glucose values (n=938,922) | 149.89 (34.32) | 147.96 (32.92)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.179, ANOVA — P-value is for Baseline mean fasting blood glucose; ANOVA with treatment, country, TZD use and sulfo use in model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for mean fasting blood glucose; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.700, ANOVA — P-value is for Baseline AM 2-hour postprandial BG; ANOVA with treatment, country, TZD use and sulfo use in model
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.016, ANCOVA — P-value for AM 2-hour postprandial blood glucose; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.971, ANOVA — P-value is for Baseline midday premeal BG; ANOVA with treatment, country, TZD use and sulfo use in model
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Midday premeal blood glucose (BG); Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.759, ANOVA — P-value is for Baseline midday 2-hour postprandial BG; ANOVA with treatment, country, TZD use and sulfo use in model
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.514, ANCOVA — P-value Midday 2-hour postprandial BG; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.321, ANOVA — P-value is for Baseline evening pre-meal BG; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.161, ANCOVA — P-value for Evening pre-meal blood glucose; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 11: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.297, ANOVA — P-value is for Baseline evening 2hour postprandial; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 12: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value Evening 2-hour postprandial BG; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 13: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.199, ANOVA — P-value is for Baseline 3 AM blood glucose; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 14: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.693, ANCOVA — P-value is for 3 AM blood glucose; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 15: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.021, ANOVA — P-value is for Baseline AM 2-hour BG excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 16: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for AM 2-hour blood glucose excursion; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 17: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.567, ANOVA — P-value is for Baseline midday 2-hour BG excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 18: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value is for Midday 2-hour blood glucose excursion; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 19: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.994, ANOVA — P-value is for Baseline PM 2-hour BG excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 20: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for PM 2-hour blood glucose excursion; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 21: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.436, ANOVA — P-value is for Baseline mean all meal time excursions; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 22: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Mean of all meal time excursions; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 23: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.628, ANOVA — P-value is for Baseline mean all 2hour PP BG; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 24: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Mean of all 2-hour postprandial BG; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 25: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.677, ANOVA — P-value is for Baseline AM/PM 2-hour postprandial BG; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 26: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for AM/PM 2-hour postprandial BG; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 27: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.364, ANOVA — P-value is for Baseline mean all premeal BG; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 28: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.055, ANCOVA — P-value is for Mean of all premeal blood glucose; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 29: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.165, ANOVA — P-value is for Baseline AM/PM 2-hour BG excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 30: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for AM/PM 2-hour blood glucose excursion; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 31: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.464, ANOVA — P-value is for Baseline mean of all BG values; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 32: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.305, ANCOVA — P-value is for Mean of all blood glucose values; Response = Treatment + Baseline + Country + TZD use + sulfo use

8. Secondary Outcome: INITIATION: Change From Baseline to Endpoint in 1,5 Anhydroglucitol (1,5 AG)
Time Frame: Baseline (Initiation), Endpoint (Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 942 | 925
micrograms per milliliter (ug/mL) | 4.61 (4.85) | 5.25 (4.85)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA model with treatment, baseline, country, TZD use, and sulfo use

9. Secondary Outcome: INITIATION: Incremental Change From Baseline in Body Weight
Time Frame: Baseline (Initiation), Weeks 6, 12, 18, 24, Endpoint (LOCF)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Groups:
- Insulin Gargine: Insulin glargine for 24 weeks.
Arm/Group | Insulin Gargine | Lispro Low Mix
Number analyzed (Participants) | 1016 | 1008
kilograms (kg)
  Change from baseline at Week 6 (n=1008,995) | 0.97 (2.48) | 1.66 (2.29)
  Change from baseline at Week 12 (n=970, 960) | 1.60 (3.41) | 2.63 (3.16)
  Change from baseline at Week 18 (n=943,927) | 2.24 (3.65) | 3.44 (3.65)
  Change from baseline at Week 24 (n=925,911) | 2.59 (4.09) | 3.76 (4.00)
  Change from baseline at endpoint (n=1016,1008) | 2.45 (4.02) | 3.60 (3.99)
Statistical Analysis 1: Comparison: Insulin Gargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for change from baseline at Week 6; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 2: Comparison: Insulin Gargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for change from baseline at Week 12; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 3: Comparison: Insulin Gargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for change from baseline at Week 18; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 4: Comparison: Insulin Gargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for change from baseline at Week 24; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 5: Comparison: Insulin Gargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for change from baseline at endpoint; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use

10. Secondary Outcome: INITIATION: Body Weight
Time Frame: Baseline (Initiation), Weeks 6, 12, 18, 24, Endpoint (LOCF)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 1046 | 1044
kilograms
  Actual weight at Baseline (n=1046,1044) | 88.23 (20.78) | 88.84 (20.97)
  Actual weight at Week 6 (n=1008,995) | 89.24 (20.88) | 90.63 (20.94)
  Actual weight at Week 12 (n=970,960) | 89.80 (20.96) | 91.79 (21.16)
  Actual weight at Week 18 (n=943,927) | 90.33 (21.17) | 92.46 (21.27)
  Actual weight at Week 24 (n=925,911) | 90.78 (21.46) | 92.63 (21.23)
  Actual weight Endpoint (n=1016,1008) | 90.74 (21.36) | 92.67 (21.19)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.497, ANOVA — P-value for Actual weight at baseline; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Actual weight at Week 6; Response = Treatment + Baseline + Country + TZD use + sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value for Actual weight at Week 12; Response = Treatment + Baseline + Country + TZD use + Sulfo use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Actual weight at Week 18; Response = Treatment + Baseline + Country + TZD use + Sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Actual weight at Week 24; Response = Treatment + Baseline + Country + TZD use + Sulfo use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-value is for Actual weight at Endpoint; Response = Treatment + Baseline + Country + TZD use + Sulfo use

11. Secondary Outcome: INITIATION: Percentage of Participants With Self-reported Hypoglycemic Episodes
Description: Hypoglycemia = any time participant feels/person observes that the participant is experiencing a sign/symptom they associate with hypoglycemia (such as hunger, dizziness, shakiness, light-headedness, sweating, irritability, headache, fast heart beat, confusion, etc) or a glucose measurement ≤70 mg/dL (≤3.9 mmol/L). Severe hypoglycemia = participant requires assistance. Qualified medical staff instructed the participants about the signs and symptoms of hypoglycemia.
Time Frame: Baseline (Initiation), Endpoint (Week 24), Overall (sum of frequencies of hypoglycemic episodes after baseline ([Week 0]).
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 1024 | 1026
percentage of participants
  Hypoglycemic episodes endpoint | 51.8 | 57.1
  Overall hypoglycemic episodes | 76.7 | 80.5
  Nocturnal hypoglycemic episodes endpoint | 34.3 | 33.9
  Nocturnal hypoglycemic episodes overall | 58.4 | 59.6
  Severe hypoglycemic episodes endpoint | 0.2 | 0.6
  Severe hypoglycemic episodes overall | 1.2 | 2.1
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel — P-value is for Hypoglycemic episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.037, Cochran-Mantel-Haenszel — P-value is for Overall hypoglycemic episodes; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.834, Cochran-Mantel-Haenszel — P-value is for Nocturnal hypoglycemic episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.585, Cochran-Mantel-Haenszel — P-value is for Nocturnal hypoglycemic episodes overall; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.241, Cochran-Mantel-Haenszel — P-value is for Severe hypoglycemic episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.080, Cochran-Mantel-Haenszel — P-value is for Severe hypoglycemic episodes overall. Initiation phase and maintenance phase are included; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use

12. Secondary Outcome: INITIATION: Rate of Self-reported Hypoglycemic Episodes
Description: Hypoglycemia = participant feels/person observes, that participant is experiencing a sign/symptom they associate with hypoglycemia (such as hunger, dizziness, shakiness, light-headedness, sweating, irritability, headache, fast heart beat, confusion, etc) or glucose measurement ≤70 mg/dL (≤3.9 mmol/L). Severe hypoglycemia = participant requires assistance. Qualified medical staff instructed the participants about the signs and symptoms of hypoglycemia.
Time Frame: Endpoint (Initiation: Week 24), Overall (incidence of hypoglycemic episodes after baseline [Week 0])
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Episodes/participant/year
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 1024 | 1026
Episodes/participant/year
  Nocturnal episodes Endpoint | 11.42 (25.31) | 8.86 (19.27)
  Nocturnal episodes Overall | 9.80 (17.50) | 9.22 (16.66)
  Severe episodes Endpoint | 0.02 (0.38) | 0.09 (0.10)
  Severe episodes Overall | 0.03 (0.31) | 0.10 (1.61)
  Hypoglycemia episodes Endpoint | 20.28 (38.25) | 24.96 (39.45)
  Hypoglycemia episodes Overall | 18.14 (28.05) | 25.49 (36.04)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.009, ANOVA — P-value is for Nocturnal episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.420, ANOVA — P-value is for Nocturnal episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.165, ANOVA — P-value is for Severe episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.167, ANOVA — P-value is for Severe episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.006, ANOVA — P-value is for Hypoglycemia episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Hypoglycemia episodes Overall; Response = Treatment + Country + TZD use + Sulfo use

13. Secondary Outcome: INITIATION: Insulin Dose
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, Endpoint (LOCF)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 1029 | 1036
units/kg/day
  Week 1 (n=994,1001) | 0.13 (0.04) | 0.24 (0.07)
  Week 2 (n=991, 987) | 0.18 (0.07) | 0.28 (0.09)
  Week 3 (n=990,968) | 0.23 (0.09) | 0.32 (0.10)
  Week 4 (n=971,958) | 0.26 (0.11) | 0.35 (0.12)
  Week 5 (n=958,930) | 0.30 (0.14) | 0.38 (0.14)
  Week 6 (n=998,1023) | 0.32 (0.15) | 0.39 (0.15)
  Week 8 (n=949,933) | 0.34 (0.17) | 0.42 (0.17)
  Week 10 (n=925,916) | 0.37 (0.19) | 0.44 (0.18)
  Week 12 (n=970,972) | 0.38 (0.20) | 0.45 (0.19)
  Week 18 (n=943,943) | 0.39 (0.22) | 0.46 (0.21)
  Week 24 (n=915,920) | 0.41 (0.23) | 0.48 (0.23)
  Endpoint (n=1029,1036) | 0.40 (0.23) | 0.47 (0.23)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 1; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 2; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 3; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 4; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 5; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 6; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 8; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 10; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 12; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.001, ANOVA — P-value is for Week 18; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 11: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 24; ANOVA with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 12: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Endpoint; ANOVA with treatment, country, TZD use, and sulfo use in the model

14. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - Age
Description: Comparison of age at baseline between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 927 | 906
years | 58.21 (9.31) | 55.85 (9.99)
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model

15. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - Origin
Description: Comparison of origin at baseline between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 927 | 906
participants
  Caucasian | 680 | 521
  African Descent | 50 | 44
  East/Southeast Asian | 11 | 28
  Hispanic | 96 | 102
  Other | 20 | 36
  Western Asian | 70 | 175
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is overall; Cochran-Mantel-Haenszel test stratified by country, TZD use, and Sulfo use

16. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: Comparison of HOMA-IR (surrogate markers of insulin resistance calculated from fasting insulin and glucose) at baseline between those participants who met their goal at Week 24 and those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%). HOMA-IR = fasting insulin (milliunits per milliliter) * fasting plasma glucose (millimoles per liter) / 22.5.
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 877 | 859
units on a scale | 4.44 (3.73) | 5.45 (5.58)
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model

17. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - HbA1c
Description: Comparison of baseline HbA1c between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 915 | 885
percent glycosylated hemoglobin | 8.66 (1.13) | 9.40 (1.25)
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with met goal/did not meet goal, country, TZD use and Sulfo use in model

18. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - Baseline HbA1c Percentage Group
Description: Comparison of baseline HbA1c percentage group (<8.5,>=8.5) between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 915 | 885
participants
  <8.5% HbA1c | 464 | 220
  >=8.5% HbA1c | 451 | 665
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is overall; Cochran-Mantel-Haenszel test stratified by country, TZD use, and sulfo use

19. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - 1,5 AG
Description: Comparison of 1,5 AG between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 916 | 889
micrograms per milliliter (ug/mL) | 5.74 (4.37) | 4.28 (3.64)
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model

20. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal at Week 24 - Pre Meals Blood Glucose, Post Meals Blood Glucose, Average of All Blood Glucose, and Fasting Blood Glucose
Description: Comparison of pre meals blood glucose, post meals blood glucose, average of all blood glucose, and fasting blood glucose between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 894 | 866
milligrams per deciliter (mg/dL)
  Pre Meals Blood Glucose (n=892,866) | 190.47 (49.67) | 209.86 (59.08)
  Post Meals Blood Glucose (n=891,865) | 228.87 (54.58) | 252.90 (60.85)
  Average of All Blood Glucose (n=894,866) | 206.43 (50.05) | 227.77 (57.04)
  Fasting Blood Glucose (n=891,864) | 189.04 (48.73) | 201.22 (57.41)
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Pre Meals Blood Glucose; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Post Meals Blood Glucose; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model
Statistical Analysis 3: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Average of All Blood Glucose; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model
Statistical Analysis 4: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Fasting Blood Glucose; ANOVA with met goal/did not meet goal, country, TZD use, and sulfo use in model

21. Secondary Outcome: INITIATION: Participant Demographics of Participants Who Did Versus Did Not Achieve HbA1c Goal - Oral Diabetes Medication at Baseline
Description: Comparison of oral diabetes medication at baseline between those participants who met their goal at Week 24 versus those who did not meet their goal at Week 24 (goal HbA1c ≤7.0%).
Time Frame: Endpoint (Initiation: Week 24)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Met Goal | Did Not Meet Goal
Number analyzed (Participants) | 917 | 901
participants
  Sulfonylurea/Metformin | 563 | 631
  TZD/Metformin | 95 | 35
  Sulfonylurea/TZD | 51 | 51
  Patients with 3 drugs (Sulfonylurea/TZD/Metformin) | 208 | 184
Statistical Analysis 1: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/Metformin; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 2: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value is for TZD/Metformin; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 3: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p = 0.969, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/TZD; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 4: Comparison: Met Goal vs Did Not Meet Goal; Test type: Superiority or Other; p = 0.225, Cochran-Mantel-Haenszel — P-value is for Patients with 3 drugs (Sulfonylurea/TZD/Metformin); Cochran-Mantel-Haenszel test stratified by country only

22. Secondary Outcome: MAINTENANCE: HbA1c at Specified Visits and Endpoint
Time Frame: Baseline (Week 0), Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, Endpoint (LOCF) (up to 2.5 years)
Population: Last observation carried forward (LOCF) method was performed on the intent-to-treat (ITT) population who had at least 1 post-baseline assessment. Maintenance baseline: Week 24.
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Groups:
- Insulin Glargine: Initiation Phase: Insulin glargine for 24 weeks. Maintenance Phase: Up to an additional 2 years of insulin glargine if glycosylated hemoglobin (HbA1c) less than or equal to 7.0 at 24 weeks.
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 418 | 471
percent glycosylated hemoglobin
  Week 0 (n=415,464) | 8.59 (1.08) | 8.69 (1.16)
  Week 12 (n=412,465) | 6.82 (0.56) | 6.75 (1.16)
  Week 24 (n=418,471) | 6.49 (0.40) | 6.49 (0.42)
  Week 36 (n=403,460) | 6.72 (0.60) | 6.71 (0.61)
  Week 48 (n=395,443) | 6.85 (0.70) | 6.80 (0.70)
  Week 60 (n=332,403) | 6.85 (0.63) | 6.83 (0.63)
  Week 72 (n=305,363) | 6.80 (0.68) | 6.79 (0.66)
  Week 84 (n=268,312) | 6.79 (0.60) | 6.74 (0.60)
  Week 96 (n=242,291) | 6.85 (0.64) | 6.73 (0.60)
  Week 108 (n=219,257) | 6.83 (0.63) | 6.72 (0.56)
  Week 120 (n=204,240) | 6.87 (0.65) | 6.75 (0.60)
  Endpoint (n=414,470) | 7.20 (0.82) | 7.10 (0.81)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.204, ANOVA — P-value is for Week 0; ANCOVA used with treatment, country, TZD use, and sulfo use in the model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is for Week 12; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.657, ANCOVA — P-value is for Week 24; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.595, ANCOVA — P-value is for Week 36; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.142, ANCOVA — P-value for Week 48; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.551, ANCOVA — P-value for Week 60; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.779, ANCOVA — P-value is for Week 72; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.175, ANCOVA — P-value is for Week 84; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.018, ANCOVA — P-value for Week 96; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.047, ANCOVA — P-value is for Week 108; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 11: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.027, ANCOVA — P-value is for Week 120; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model
Statistical Analysis 12: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value is for Endpoint; ANCOVA used with treatment, baseline HbA1c, country, TZD use, and sulfo use in the model

23. Secondary Outcome: MAINTENANCE: 7-point SMPG Profiles and Postprandial Excursions
Description: as for outcome 7
Time Frame: Baseline (Maintenance: Week 24), Endpoint (LOCF) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 405 | 457
mg/dL
  Baseline mean fasting blood glucose (n=403,456) | 190.90 (48.90) | 187.12 (48.16)
  Endpoint mean fasting blood glucose (n=372,426) | 119.50 (29.04) | 127.92 (32.90)
  Baseline AM 2-hour (hr) postprandial (n=398,455) | 243.62 (58.58) | 243.55 (61.38)
  Endpoint AM 2-hour postprandial (n=368,426) | 164.94 (44.29) | 161.37 (44.66)
  Baseline midday premeal blood glucose (n=400,454) | 193.21 (61.66) | 192.02 (60.21)
  Endpoint midday premeal blood glucose (n=370,425) | 132.25 (38.28) | 126.42 (37.84)
  Baseline midday 2hr postprandial (n=397,456) | 217.67 (61.90) | 218.54 (60.65)
  Endpoint midday 2hr postprandial (n=370,424) | 159.81 (42.21) | 158.58 (40.00)
  Baseline PM pre-meal blood glucose (n=402,455) | 190.06 (57.83) | 187.92 (56.68)
  Endpoint PM pre-meal blood glucose (n=371,425) | 131.58 (37.22) | 133.15 (37.30)
  Baseline PM 2hr postprandial (n=399,455) | 223.83 (62.70) | 223.02 (60.64)
  Endpoint PM 2hr postprandial (n=369,425) | 167.66 (43.81) | 156.48 (44.10)
  Baseline 3AM blood glucose (n=393,450) | 189.36 (59.87) | 183.18 (57.15)
  Endpoint 3AM blood glucose (n=363,419) | 126.05 (34.33) | 123.43 (35.37)
  Baseline AM 2hr excursion (n=397,455) | 52.63 (44.06) | 56.96 (45.40)
  Endpoint AM 2hr excursion (n=368,426) | 45.69 (39.41) | 33.61 (38.67)
  Baseline midday 2hr excursion (n=395,452) | 25.13 (46.67) | 27.02 (43.17)
  Endpoint midday 2hr excursion (n=370,423) | 27.78 (37.38) | 32.03 (38.64)
  Baseline PM 2hr excursion (n=398,453) | 33.87 (42.37) | 34.78 (44.40)
  Endpoint PM 2hr excursion (n=369,424) | 36.24 (37.55) | 23.45 (41.99)
  Baseline mean all meal time excursions (n=402,455) | 37.36 (27.26) | 39.65 (25.60)
  Endpoint mean all meal time excursions (n=370,426) | 36.32 (26.25) | 29.81 (27.04)
  Baseline mean of all 2hr postprandial (n=402,457) | 228.52 (54.01) | 228.39 (53.63)
  Endpoint mean of all 2hr postprandial (n=370,426) | 164.17 (36.30) | 158.91 (36.07)
  Baseline mean all premeal (n=404,456) | 191.46 (50.02) | 188.95 (48.34)
  Endpoint mean all premeal (n=372,426) | 127.61 (28.40) | 129.16 (29.41)
  Baseline combined AM/PM 2hr postprandial (402,457) | 233.82 (55.31) | 233.25 (55.06)
  Endpoint combined AM/PM 2hr postprandial (370,426) | 166.34 (38.28) | 158.97 (38.59)
  Baseline AM/PM 2hr postprandial excursion (402,455 | 43.46 (32.72) | 45.80 (33.80)
  Endpoint AM/PM 2hr postprandial excursion (370,426 | 40.76 (32.01) | 28.69 (31.08)
  Baseline mean all blood glucose values (n=405,457) | 207.01 (49.91) | 205.17 (48.86)
  Endpoint mean all blood glucose values (n=372,426) | 142.94 (29.16) | 141.01 (28.97)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.218, ANOVA — P-value for Baseline mean fasting blood glucose; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint mean fasting blood glucose; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.897, ANOVA — P-value is for Baseline AM 2-hour (hr) postprandial; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.138, ANCOVA — P-value is for Endpoint AM 2-hour postprandial; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.867, ANOVA — P-value is for Baseline midday premeal blood glucose; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.031, ANCOVA — P-value is for Endpoint midday premeal blood; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.792, ANOVA — P-value is for Baseline midday 2hr postprandial; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.510, ANCOVA — P-value is for Endpoint midday 2hr postprandial; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.535, ANOVA — P-value is for Baseline PM pre-meal blood glucose; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.517, ANCOVA — P-value is for Endpoint PM pre-meal blood glucose; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 11: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.869, ANOVA — P-value is for Baseline PM 2hr postprandial; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 12: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint PM 2hr postprandial; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 13: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.164, ANOVA — P-value is for Baseline 3AM blood glucose; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 14: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.234, ANCOVA — P-value is for Endpoint 3AM blood glucose; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 15: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.175, ANOVA — P-value is for Baseline AM 2hr excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 16: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint AM 2hr excursion; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 17: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.589, ANOVA — P-value is for Baseline midday 2hr excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 18: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.161, ANCOVA — P-value is for Endpoint midday 2hr excursion; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 19: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.674, ANOVA — P-value is for Baseline PM 2hr excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 20: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint PM 2hr excursion; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 21: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.201, ANOVA — P-value is for Baseline mean all meal time excursions; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 22: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint mean all meal time excursions; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 23: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.956, ANOVA — P-value is for Baseline mean of all 2hr postprandial; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 24: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.019, ANCOVA — P-value is for Endpoint mean of all 2hr postprandial; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 25: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.445, ANOVA — P-value is for Baseline mean all premeal; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 26: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.371, ANOVA — P-value is for Endpoint mean all premeal; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 27: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.848, ANOVA — P-value is for Baseline combined AM/PM 2hr postprandial; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 28: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is for Endpoint combined AM/PM 2hr postprandial; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 29: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.281, ANOVA — P-value is for Baseline AM/PM 2hr postprandial excursion; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 30: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint AM/PM 2hr postprandial excursion; Response = Treatment + Baseline + Country + TZD + Sulfo use
Statistical Analysis 31: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.588, ANOVA — P-value is for Baseline mean all blood glucose values; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 32: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.217, ANCOVA — P-value is for Endpoint mean all blood glucose values; Response = Treatment + Baseline + Country + TZD + Sulfo use

24. Secondary Outcome: MAINTENANCE: Rate of Increase in HbA1c
Description: Rate of increase: HbA1c change/time period (month).
Time Frame: Endpoint (LOCF) (Maintenance: up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: HbA1c percent increase per month
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 412 | 469
HbA1c percent increase per month | 0.06 (0.08) | 0.05 (0.09)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.300, ANCOVA; ANCOVA used with treatment, Baseline HbA1c, country, TZD use, and sulfo use in the model

25. Secondary Outcome: MAINTENANCE: Percentage of Participants With HbA1c < or = 7.0%, HbA1c <7.0, and HbA1c < or = 6.5%
Time Frame: Endpoint (LOCF) (Maintenance: up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 414 | 470
percentage of participants
  <=7.0% | 44.9 | 49.1
  <7.0% | 40.1 | 45.1
  <=6.5% | 23.7 | 26.4
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.134, Cochran-Mantel-Haenszel — P-value for <=7.0%; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.089, Cochran-Mantel-Haenszel — P-value is for <7.0%; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.235, Cochran-Mantel-Haenszel — P-value is for <=6.5%; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use

26. Secondary Outcome: MAINTENANCE: Incremental Change From Baseline in Body Weight
Time Frame: Baseline (Week 0), Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 419 | 473
kilograms
  Baseline (n=419,473) | 90.56 (20.12) | 88.62 (19.05)
  Change from baseline at Week 24 (n=417,470) | 2.05 (3.79) | 3.68 (3.89)
  Change from baseline at Week 36 (n=411,465) | 2.71 (4.22) | 4.56 (4.44)
  Change from baseline at Week 48 (n=399,460) | 3.08 (4.46) | 4.82 (4.81)
  Change from baseline at Week 60 (n=362,414) | 3.33 (4.76) | 5.13 (5.22)
  Change from baseline at Week 72 (n=315,372) | 3.12 (5.15) | 5.40 (5.72)
  Change from baseline at Week 84 (n=281,327) | 3.16 (5.20) | 5.84 (5.87)
  Change from baseline at Week 96 (n=248,297) | 3.11 (5.35) | 5.60 (5.68)
  Change from baseline at Week 108 (n=228,268) | 3.48 (5.65) | 5.57 (5.66)
  Change from baseline at Week 120 (n=204,253) | 3.71 (5.47) | 5.48 (5.88)
  Change from baseline at Endpoint (n=414,470) | 3.65 (5.60) | 5.40 (5.83)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 24; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 36; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 48; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 60; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 72; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 84; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 96; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Week 108; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is for Change from baseline at Week 120; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Change from baseline at Endpoint; Model: Response = Treatment + Baseline + Country + TZD use + sulfonylurea use

27. Secondary Outcome: MAINTENANCE: Body Weight
Time Frame: Baseline (Week 0), Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 419 | 473
kilograms
  Baseline (n=419,473) | 90.56 (20.12) | 88.62 (19.05)
  Week 24 (n=417, 470) | 92.64 (20.53) | 92.35 (19.10)
  Week 36 (n=411, 465) | 93.13 (20.68) | 93.24 (19.38)
  Week 48 (n=399,460) | 93.23 (20.53) | 93.57 (19.41)
  Week 60 (n=362,414) | 93.17 (20.60) | 94.57 (19.62)
  Week 72 (n=315,372) | 93.62 (20.40) | 95.50 (19.63)
  Week 84 (n=281,327) | 93.46 (20.56) | 95.63 (19.78)
  Week 96 (n=248, 297) | 93.33 (20.14) | 95.34 (19.50)
  Week 108 (n=228,268) | 93.39 (20.23) | 95.07 (19.61)
  Week 120 (n=204,253) | 93.99 (20.22) | 94.82 (19.62)
  Endpoint (n=414,470) | 94.14 (21.04) | 94.01 (19.92)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.128, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 36; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 48; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 60; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 72; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 84; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 96; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Week 108; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is for Week 120; Response = Treatment + Baseline + Country + TZD use + Sulfo Use
Statistical Analysis 11: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use + Sulfo Use

28. Secondary Outcome: MAINTENANCE: Insulin Dose
Time Frame: Weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 418 | 473
units/kg/day
  Week 24 (n=418,473) | 0.36 (0.19) | 0.43 (0.19)
  Week 36 (n=415,470) | 0.36 (0.19) | 0.44 (0.20)
  Week 48 (n=407,464) | 0.37 (0.20) | 0.44 (0.20)
  Week 60 (n=364,419) | 0.37 (0.19) | 0.44 (0.19)
  Week 72 (n=317,374) | 0.37 (0.20) | 0.44 (0.20)
  Week 84 (n=284,334) | 0.36 (0.20) | 0.44 (0.21)
  Week 96 (n=251,303) | 0.37 (0.21) | 0.44 (0.21)
  Week 108 (n=233,273) | 0.36 (0.20) | 0.43 (0.21)
  Week 120 (n=205,254) | 0.36 (0.20) | 0.44 (0.21)
  Endpoint (n=416,472) | 0.37 (0.21) | 0.45 (0.21)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 24; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 36; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 48; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 60; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 72; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 84; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 7: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 96; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 8: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 108; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 9: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Week 120; Model: Treatment + Country + TZD use + sulfonylurea use
Statistical Analysis 10: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p < 0.001, ANOVA — P-value is for Endpoint; Model: Treatment + Country + TZD use + sulfonylurea use

29. Secondary Outcome: MAINTENANCE: Percentage of Participants With Self-reported Hypoglycemic Episodes
Description: Hypoglycemia = participant feels/person observes that the participant is experiencing a sign/symptom they associate with hypoglycemia (such as hunger, dizziness, shakiness, light-headedness, sweating, irritability, headache, fast heart beat, confusion, etc) or a glucose measurement ≤70 mg/dL (≤3.9 mmol/L). Severe hypoglycemia = participant requires assistance. Qualified medical staff instructed the participants about the signs and symptoms of hypoglycemia.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years), Overall (incidence of hypoglycemic episodes after baseline (Week 0)
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 419 | 473
percentage of participants
  Overall hypoglycemic episodes endpoint (n=415,471) | 45.3 | 49.9
  Overall hypoglycemic episodes (n=419,473) | 94.0 | 97.9
  Nocturnal episodes endpoint (n=415,471) | 30.4 | 28.9
  Nocturnal episodes overall (n=419,473) | 81.1 | 84.4
  Severe episodes endpoint (n=415,471) | 0.5 | 0.6
  Severe episodes overall (n=419,473) | 2.9 | 4.2
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.370, Cochran-Mantel-Haenszel — P-value is for Overall hypoglycemic episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — P-Value for Overall hypoglycemia episodes; Controlling for country, TZD use, and sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.397, Cochran-Mantel-Haenszel — P-value is for Nocturnal episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.253, Cochran-Mantel-Haenszel — P-value is for Nocturnal episodes overall; Controlling for country, TZD use, and sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.893, Cochran-Mantel-Haenszel — P-value is for Severe episodes endpoint; Controlling for country, TZD use, and sulfo use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.391, Cochran-Mantel-Haenszel — P-value is for Severe episodes overall; Cochran-Mantel-Haenszel statistic controlling for country, TZD use, and sulfo use

30. Secondary Outcome: MAINTENANCE: Rate of Self-reported Hypoglycemic Episodes
Description: as for outcome 29
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years), Overall (incidence of hypoglycemic episodes after baseline [Week 0])
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: episodes/participant/year
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 415 | 471
episodes/participant/year
  Hypoglycemia episodes Endpoint | 16.41 (34.78) | 18.56 (35.50)
  Hypoglycemia episodes Overall | 21.80 (26.77) | 26.08 (31.69)
  Nocturnal episodes Endpoint | 7.70 (19.36) | 5.86 (15.96)
  Nocturnal episodes Overall | 9.77 (15.01) | 8.02 (13.49)
  Severe episodes Endpoint | 0.23 (4.43) | 0.03 (0.46)
  Severe episodes Overall | 0.12 (2.12) | 0.03 (0.21)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.497, ANOVA — P-value for Hypoglycemia episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.071, ANOVA — P-value is for Hypoglycemia episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.065, ANOVA — P-value is for Nocturnal episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 4: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.021, ANOVA — P-value is for Nocturnal episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 5: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.200, ANOVA — P-value is for Severe episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 6: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.208, ANOVA — P-value is for Severe episodes Overall; Response = Treatment + Country + TZD use + Sulfo use

31. Secondary Outcome: MAINTENANCE: Change From Baseline in 1,5-Anhydroglucitol
Time Frame: Baseline (Maintenance: Week 24), Endpoint (LOCF) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 372 | 428
ug/dL
  Baseline | 5.66 (4.34) | 5.87 (4.51)
  Endpoint | 10.48 (6.26) | 11.71 (6.44)
  Change | 4.82 (5.28) | 5.84 (5.19)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is for Change; ANCOVA model with treatment, baseline, country, TZD use and sulfo use

32. Secondary Outcome: MAINTENANCE: Change From Baseline to Endpoint in HbA1c
Time Frame: Baseline (Week 0), Week 24, Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Insulin Glargine | Lispro Low Mix
Number analyzed (Participants) | 415 | 469
percent glycosylated hemoglobin
  Baseline at Week 0 (n=415,464) | 8.59 (1.08) | 8.69 (1.16)
  Change from baseline to endpoint (n=409,462) | -1.38 (1.18) | -1.59 (1.22)
  Change Week 24 to Week 120 endpoint (n=412,469) | 0.71 (0.11) | 0.61 (0.75)
Statistical Analysis 1: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.204, ANOVA — P-value is for Baseline at Week 0; ANOVA used with treatment, country, TZD use and Sulfo use in the model
Statistical Analysis 2: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.017, ANCOVA — P-Value is for Change from baseline to endpoint; ANCOVA used with treatment, Baseline HbA1c, country, TZD use and sulfo use in the model
Statistical Analysis 3: Comparison: Insulin Glargine vs Lispro Low Mix; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value is for Change Week 24 to Week 120 endpoint; ANCOVA used with treatment, Baseline HbA1c, country, TZD use and sulfo use in the model

33. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - Duration of Diabetes
Description: Comparison of duration of diabetes at baseline between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 147 | 272
years | 8.44 (4.92) | 9.70 (6.12)
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.036, ANOVA; ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

34. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - Duration of Diabetes
Description: Comparison of duration of diabetes at baseline between those participants taking lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 202 | 271
years | 9.42 (6.24) | 9.87 (6.38)
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.708, ANOVA; From ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

35. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - Duration of Diabetes Group
Description: Comparison of duration of diabetes group (<10, 10-<20, >=20 years) at baseline between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 147 | 272
participants
  Less than 10 years | 96 | 152
  10 years to less than 20 years | 45 | 94
  20 or more years | 6 | 26
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by country, TZD use, and Sulfo use

36. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - Duration of Diabetes Group
Description: Comparison of duration of diabetes group (<10, 10-<20, >=20 years) at baseline between those participants taking Lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 202 | 271
participants
  <10 years | 112 | 148
  10 to <20 years | 78 | 97
  >=20 years | 12 | 26
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.738, Cochran-Mantel-Haenszel; Stratified by country, TZD use, and sulfo use

37. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - Baseline HbA1c
Description: Comparison of baseline HbA1c between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 143 | 270
percent glycosylated hemoglobin | 8.27 (0.94) | 8.77 (1.11)
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p < 0.001, ANOVA; ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

38. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - Baseline HbA1c
Description: Comparison of baseline HbA1c between those participants taking Lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 198 | 268
percent glycosylated hemoglobin | 8.54 (1.13) | 8.80 (1.17)
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.043, ANOVA; ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

39. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - Baseline HbA1c Group
Description: Comparison of baseline HbA1c group (<8.5,>=8.5) between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 143 | 270
participants
  Less than 8.5% HbA1c | 97 | 121
  >=8.5% HbA1c | 46 | 149
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by country, TZD use, and sulfo use

40. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - Baseline HbA1c Group
Description: Comparison of baseline HbA1c group (<8.5,>=8.5) between those participants taking Lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 198 | 268
participants
  Less than 8.5 | 110 | 121
  8.5 or more | 88 | 147
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.032, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by country, TZD use, and sulfo use

41. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - Oral Diabetes Medicine at Baseline
Description: Comparison of oral diabetes medication at baseline between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 144 | 269
participants
  Sulfonylurea/TZD | 16 | 13
  Sulfonylurea/metformin | 73 | 175
  Metformin/TZD | 22 | 22
  Sulfonylurea/metformin/TZD | 33 | 59
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.037, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/TZD; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 2: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/metformin; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 3: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.132, Cochran-Mantel-Haenszel — P-value is for Metformin/TZD; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 4: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.849, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/metformin/TZD; Cochran-Mantel-Haenszel test stratified by country only

42. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - Oral Diabetes Medicine at Baseline
Description: Comparison of oral diabetes medication at baseline between those participants taking Lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Number; unit: participants
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 199 | 270
participants
  Sulfonylurea/TZD | 14 | 5
  Sulfonylurea/metformin | 115 | 185
  Metformin/TZD | 25 | 21
  Sulfonylurea/metformin/TZD | 45 | 59
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/TZD; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 2: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/metformin; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 3: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.258, Cochran-Mantel-Haenszel — P-value is for Metformin/TZD; Cochran-Mantel-Haenszel test stratified by country only
Statistical Analysis 4: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.848, Cochran-Mantel-Haenszel — P-value is for Sulfonylurea/metformin/TZD; Cochran-Mantel-Haenszel test stratified by country only

43. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - 1,5 AG
Description: Comparison of baseline 1,5 AG between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 146 | 271
ug/mL | 6.29 (4.60) | 5.39 (4.22)
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.004, ANOVA; ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

44. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - 1,5 AG
Description: Comparison of baseline 1,5 AG between those participants taking Lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 199 | 265
ug/ml | 5.93 (4.17) | 5.73 (4.64)
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.553, ANOVA; From ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

45. Secondary Outcome: MAINTENANCE: Participant Demographics of Insulin Glargine Participants Who Did Versus Did Not Maintain HbA1c Goal - Mean of Post Meals Blood Glucose and Average of All Blood Glucose
Description: Comparison of baseline mean of post meals blood glucose and average of all blood glucose between those participants taking insulin glargine that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glargine Participants Who Maintained Goal | Insulin Glargine Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 141 | 264
mg/dL
  Mean of post meals blood glucose (n=141,261) | 219.28 (51.23) | 233.51 (54.90)
  Average of all blood glucose (n=141,264) | 200.60 (48.07) | 210.44 (50.63)
Statistical Analysis 1: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.010, ANOVA — P-value is for Mean of all post meals blood glucose; ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Insulin Glargine Participants Who Maintained Goal vs Insulin Glargine Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.035, ANOVA — P-value is for Average of all blood glucose; ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

46. Secondary Outcome: MAINTENANCE: Participant Demographics of Lispro LM Participants Who Did Versus Did Not Maintain HbA1c Goal - Mean of Post Meals Blood Glucose and Average of All Blood Glucose
Description: Comparison of baseline mean of post meals blood glucose and average of all blood glucose between those participants taking Lispro LM that maintained their HbA1c goal and those that did not. Participants who maintained goal are those who did not fail during their duration on study. Failure is defined by HbA1c > 7.0% with change >= 0.4% from most recent HbA1c that was <=7.0%.
Time Frame: Endpoint (LOCF) (Maintenance) (up to 2.5 years)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lispro LM Participants Who Maintained Goal | Lispro LM Participants Who Did Not Maintain Goal
Number analyzed (Participants) | 195 | 262
mg/dL
  Mean of post meals blood glucose | 223.98 (52.54) | 231.66 (54.30)
  Average of all blood glucose | 201.42 (48.42) | 207.96 (49.09)
Statistical Analysis 1: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.516, ANOVA — P-value is for Mean of post-meals blood glucose; From ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model
Statistical Analysis 2: Comparison: Lispro LM Participants Who Maintained Goal vs Lispro LM Participants Who Did Not Maintain Goal; Test type: Superiority or Other; p = 0.425, ANOVA — P-value is for Average of all blood glucose; From ANOVA with maintained goal/did not maintain goal, country, TZD use, and sulfo use in model

47. Secondary Outcome: ADDENDUM: Change in HbA1c From Point of Second Randomization (Addendum Baseline) to Endpoint
Time Frame: Baseline (Addendum: Week 24), Endpoint (24 weeks [Week 48])
Population: Last observation carried forward (LOCF) method was performed on the intent-to-treat (ITT) population who had at least 1 post-baseline assessment. Addendum baseline: 24 weeks: Week 48.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro LM Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Number analyzed (Participants) | 174 | 200 | 171 | 199
percent
  Baseline (n=174,200,171,199) | 8.01 (0.93) | 8.03 (0.95) | 8.00 (0.92) | 7.98 (0.95)
  Endpoint (n=160,187,159,176) | 0.19 (1.12) | 0.04 (1.06) | 0.19 (1.16) | 0.18 (1.26)
Statistical Analysis 1: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.770, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 2: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.990, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 3: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.552, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 4: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.271, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use

48. Secondary Outcome: ADDENDUM: Percentage of Participants With HbA1c < or = 7.0%, HbA1c < 7.0%, and < or = 6.5%
Time Frame: Endpoint (Addendum: 24 weeks [Week 48])
Population: as for outcome 47
Measure: Number; unit: percent of participants
Arm/Group | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro LM Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Number analyzed (Participants) | 176 | 187 | 159 | 176
percent of participants
  <=7.0% | 12.5 | 16.0 | 22.0 | 18.2
  <7.0% | 8.8 | 13.9 | 17.6 | 4.0
  <=6.5% | 4.4 | 3.7 | 5.0 | 4.0
Statistical Analysis 1: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.027, Fisher Exact — P-value is for <=7.0%
Statistical Analysis 2: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.021, Fisher Exact — P-value is for <7.0%
Statistical Analysis 3: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.799, Fisher Exact — P-value is for <=6.5%
Statistical Analysis 4: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.676, Fisher Exact — P-value is for <=7.0%
Statistical Analysis 5: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is for <7.0%
Statistical Analysis 6: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value is for <=6.5%

49. Secondary Outcome: ADDENDUM: 7-point SMPG Profiles
Description: as for outcome 7
Time Frame: Endpoint (Addendum: 24 weeks [Week 48])
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Basal Bolus Prior Lispro LM Addendum; Lispro Low Mix Prior Glargine Addendum: Following Lispro LM Initiation Phase, if HbA1c greater than 7.0 after 24 weeks, then instead of entering Maintenance Phase, they could be randomized to receive Basal Bolus therapy (combination of insulin glargine and lispro) for 24 weeks in the Intensification Addendum Phase.
Arm/Group | Basal Bolus Prior Lispro LM Addendum | Lispro Mid Mix Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum | Lispro Low Mix Prior Glargine Addendum
Number analyzed (Participants) | 152 | 161 | 183 | 187
mg/dL
  Mean fast blood glucose (BG) (n=135,150,161,178) | 145.33 (35.23) | 151.15 (37.31) | 126.22 (39.00) | 139.45 (34.92)
  AM 2-hour postprandial (PP) BG (n=135,149,160,176) | 168.71 (44.90) | 170.36 (50.25) | 170.14 (49.27) | 171.40 (46.90)
  Midday premeal blood glucose (n=135,150,161,177) | 144.08 (43.93) | 145.89 (42.61) | 144.61 (41.39) | 141.87 (43.33)
  Midday 2-hour (hr) PP BG (n=135,149,160,176)) | 165.24 (46.46) | 164.13 (42.17) | 167.45 (48.27) | 181.46 (53.34)
  PM premeal blood glucose (n=135,150,161,178) | 153.62 (41.82) | 151.96 (41.66) | 157.15 (54.22) | 153.19 (40.74)
  PM 2-hour postprandial BG (n=134,150,161,178) | 171.51 (44.42) | 172.98 (48.01) | 175.34 (53.17) | 174.94 (46.73)
  3 AM blood glucose (n=132,146,153,171) | 146.50 (40.09) | 146.30 (41.36) | 147.14 (39.99) | 139.86 (39.15)
  AM 2-hour BG excursion (n=135,149,160,176) | 23.30 (39.14) | 18.97 (46.88) | 24.35 (38.44) | 31.33 (43.27)
  Midday 2-hour BG excursion (n=135,148,160,176) | 20.71 (43.35) | 18.97 (41.40) | 23.30 (37.21) | 39.40 (46.21)
  PM 2-hour BG excursion (n=134,150,161,178) | 17.88 (38.16) | 21.14 (42.48) | 18.58 (41.86) | 21.59 (43.88)
  Mean all mealtime excursions (n=135,150,161,178) | 20.61 (28.41) | 19.64 (27.87) | 21.82 (26.09) | 30.38 (31.11)
  Mean all 2-hour PP BG (n=135,150,161,178) | 168.55 (38.92) | 169.14 (39.27) | 170.95 (42.89) | 175.61 (42.15)
  Mean all premeal blood glucose (n=135,150,161,178) | 147.68 (32.85) | 149.67 (33.20) | 149.04 (38.35) | 144.85 (32.07)
  Mean combined AM/PM 2hr PP BG (n=135,150,161,178) | 170.04 (39.98) | 171.65 (43.23) | 172.73 (45.15) | 172.88 (41.56)
  Mean AM/PM 2hr BG excursion (n=135,150,161,178) | 20.74 (30.40) | 20.06 (34.62) | 21.42 (32.09) | 26.45 (33.36)
  Mean all BG values (n=135,150,161,178) | 156.41 (33.04) | 157.52 (32.67) | 158.33 (37.89) | 157.41 (33.21)
  Baseline mean all premeals BG (n=152,161,183,187) | 149.91 (38.96) | 149.50 (34.82) | 146.64 (39.89) | 146.01 (34.80)
  Baseline mean of postmeal BG (n=152,161,182,187) | 183.82 (45.13) | 181.18 (43.49) | 186.19 (46.23) | 185.62 (41.67)
  Baseline average of all BG (n=152,161,183,187) | 164.02 (39.20) | 162.18 (35.22) | 163.19 (40.08) | 163.20 (34.69)
  Baseline fasting glucose (n=152,161,183,187) | 147.93 (39.46) | 143.99 (34.91) | 131.54 (42.16) | 131.02 (34.91)
Statistical Analysis 1: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.241, ANCOVA — P-value is for Mean fast blood glucose (BG); Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 2: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.305, ANCOVA — P-value is for AM 2-hour postprandial (PP) BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 3: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.842, ANCOVA — P-value is for Midday premeal blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 4: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.917, ANCOVA — P-value is for Midday 2-hour (hr) PP BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 5: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.648, ANCOVA — P-value is for PM premeal blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 6: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.613, ANCOVA — P-value is for PM 2-hour postprandial BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 7: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.813, ANCOVA — P-value is for 3 AM blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 8: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.953, ANCOVA — P-value is for AM 2-hour BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 9: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.933, ANCOVA — P-value is for Midday 2-hour BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 10: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.348, ANCOVA — P-value is for PM 2-hour BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 11: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.625, ANCOVA — P-value is for Mean all mealtime excursions; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 12: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.573, ANCOVA — P-value is for Mean all 2-hour PP BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 13: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.711, ANCOVA — P-value is for Mean all premeal blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 14: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.372, ANCOVA — P-value is for Mean combined AM/PM 2hr PP BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 15: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.516, ANCOVA — P-value is for Mean AM/PM 2hr BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 16: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.639, ANCOVA — P-value is for Mean all BG values; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 17: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.131, ANCOVA — P-value is for Mean fast blood glucose (BG); Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 18: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.530, ANCOVA — P-value is for AM 2-hour postprandial (PP) BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 19: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.578, ANCOVA — P-value is for Midday premeal blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 20: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is for Midday 2-hour (hr) PP BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 21: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.951, ANCOVA — P-value is for PM premeal blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 22: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.580, ANCOVA — P-value is for PM 2-hour postprandial BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 23: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.071, ANCOVA — P-value is for 3 AM blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 24: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.081, ANCOVA — P-value is for AM 2-hour BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 25: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for Midday 2-hour BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 26: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.542, ANCOVA — P-value is for PM 2-hour BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 27: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.003, ANCOVA — P-value is for Mean all mealtime excursions; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 28: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.105, ANCOVA — P-value is for Mean all 2-hour PP BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 29: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.487, ANCOVA — P-value is for Mean all premeal blood glucose; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 30: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.491, ANCOVA — P-value is for Mean combined AM/PM 2hr PP BG; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 31: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.127, ANCOVA — P-value is for Mean AM/PM 2hr BG excursion; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 32: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.861, ANCOVA — P-value is for Mean all BG values; Response = Treatment + Baseline + Country + TZD use

50. Secondary Outcome: ADDENDUM: Incremental Change From Baseline in Body Weight
Time Frame: Baseline (Addendum: Week 24), Weeks 6 (30 Weeks), 12 (36 Weeks), 24 (48 Weeks), Endpoint (LOCF)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Basal Bolus Prior Lispro LM Addendum | Lispro Mid Mix Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum | Lispro Low Mix Prior Glargine Addendum
Number analyzed (Participants) | 170 | 173 | 198 | 200
kilograms
  Baseline (n=170,173,198,200) | 91.85 (23.41) | 93.63 (24.21) | 89.25 (21.62) | 90.09 (23.45)
  Week 6 change (n=161,162,183,193) | 0.38 (2.78) | 0.28 (1.76) | 0.32 (2.15) | 0.64 (2.10)
  Week 12 change (n=150,158,173,187) | 0.43 (2.61) | 0.54 (2.36) | 0.27 (3.31) | 0.83 (2.37)
  Week 24 change (n=144,151,163,176) | 0.77 (3.01) | 0.73 (2.85) | 1.03 (3.24) | 1.51 (3.11)
  Endpoint change (n=163,169,191,198) | 0.85 (3.46) | 0.55 (2.85) | 0.86 (3.41) | 1.42 (3.03)
Statistical Analysis 1: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.745, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 2: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.467, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 3: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.575, ANCOVA — P-value is for Week 6; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 4: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.726, ANCOVA — P-value is for Week 12; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 5: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.978, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 6: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.345, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 7: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.166, ANCOVA — P-value is for Week 6; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 8: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value is for Week 12; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 9: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.199, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 10: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.098, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use

51. Secondary Outcome: ADDENDUM: Body Weight
Time Frame: Baseline (Addendum Week 24), Weeks 6 (30 weeks), 12 (36 weeks), 24 (48 weeks), Endpoint (LOCF)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Basal Bolus Prior Lispro LM Addendum | Lispro Mid Mix Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum | Lispro Low Mix Prior Glargine Addendum
Number analyzed (Participants) | 170 | 173 | 198 | 200
kilograms
  Baseline (n=170,173,198,200) | 91.85 (23.41) | 93.63 (24.21) | 89.25 (21.62) | 90.09 (23.45)
  Week 6 (n=162,163,184,193) | 91.53 (23.33) | 93.71 (24.82) | 89.66 (21.97) | 89.85 (22.50)
  Week 12 (n=151,158,174,187) | 91.59 (22.88) | 94.60 (25.08) | 89.62 (22.04) | 91.19 (23.68)
  Week 24 (n=145,151,164,176) | 91.92 (23.32) | 94.18 (24.99) | 89.80 (21.95) | 91.22 (23.30)
  Endpoint (n=164,170,192,198) | 92.40 (23.67) | 94.09 (24.65) | 90.09 (21.95) | 91.45 (23.64)
Statistical Analysis 1: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.467, ANOVA — P-value is for Baseline; ANOVA with treatment, country, and TZD use in model
Statistical Analysis 2: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.575, ANCOVA — P-value is for Week 6; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 3: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.726, ANCOVA — P-value is for Week 12; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 4: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.978, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 5: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.345, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 6: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.745, ANOVA — P-value is for Baseline; ANOVA with treatment, country, and TZD use in model
Statistical Analysis 7: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.166, ANCOVA — P-value is for Week 6; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 8: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.064, ANCOVA — P-value is for Week 12; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 9: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.199, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 10: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.098, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use

52. Secondary Outcome: ADDENDUM: Insulin Dose
Time Frame: Baseline (Addendum: Week 24), Weeks 1 (25 weeks), 2 (26 weeks), 3 (27 weeks), 4 (28 weeks), 5 (25 weeks), 6 (26 weeks), 8 (32 weeks), 10 (34 weeks), 12 (36 weeks), 24 (48 weeks), Endpoint (LOCF)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Basal Bolus Prior Lispro LM Addendum | Lispro Mid Mix Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum | Lispro Low Mix Prior Glargine Addendum
Number analyzed (Participants) | 171 | 174 | 199 | 200
units/kg/day
  Baseline (n=171,174,199,200) | 0.55 (0.26) | 0.55 (0.25) | 0.46 (0.27) | 0.46 (0.24)
  Week 1 (n=152,158,183,183) | 0.58 (0.26) | 0.57 (0.25) | 0.49 (0.27) | 0.49 (0.25)
  Week 2 (n=147,159,180,187) | 0.63 (0.29) | 0.59 (0.26) | 0.54 (0.29) | 0.53 (0.24)
  Week 3 (n=149,158,179,184) | 0.65 (0.28) | 0.64 (0.26) | 0.57 (0.28) | 0.58 (0.24)
  Week 4 (n=145,157,178,178) | 0.69 (0.29) | 0.67 (0.27) | 0.63 (0.34) | 0.61 (0.25)
  Week 5 (n=148,153,172,173) | 0.73 (0.29) | 0.70 (0.28) | 0.65 (0.34) | 0.65 (0.26)
  Week 6 (n=162,168,190,196) | 0.73 (0.29) | 0.72 (0.29) | 0.68 (0.37) | 0.66 (0.28)
  Week 8 (n=139,154,164,174) | 0.76 (0.29) | 0.75 (0.32) | 0.71 (0.38) | 0.69 (0.29)
  Week 10 (n=141,152,158,174) | 0.78 (0.31) | 0.77 (0.32) | 0.76 (0.43) | 0.73 (0.31)
  Week 12 (n=152,161,177,190) | 0.80 (0.33) | 0.79 (0.33) | 0.77 (0.42) | 0.74 (0.32)
  Week 24 (n=147,151,166,179) | 0.82 (0.35) | 0.80 (0.35) | 0.79 (0.45) | 0.76 (0.32)
  Endpoint (n=165,170,199,200) | 0.81 (0.35) | 0.79 (0.35) | 0.77 (0.43) | 0.76 (0.33)
Statistical Analysis 1: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.837, ANOVA — P-value is for Week 1; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 2: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.205, ANOVA — P-value is for Week 2; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 3: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.704, ANOVA — P-value is for Week 3; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 4: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.610, ANOVA — P-value is for Week 4; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 5: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.352, ANOVA — P-value is for Week 5; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 6: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.636, ANOVA — P-value is for Week 6; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 7: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.880, ANOVA — P-value is for Week 8; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 8: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.904, ANOVA — P-value is for Week 10; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 9: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.859, ANOVA — P-value is for Week 12; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 10: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.654, ANOVA — P-value is for Week 24; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 11: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.566, ANOVA — P-value is for Endpoint; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 12: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.926, ANOVA — P-value is for Week 1; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 13: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.902, ANOVA — P-value is for Week 2; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 14: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.766, ANOVA — P-value is for Week 3; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 15: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.449, ANOVA — P-value is for Week 4; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 16: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.797, ANOVA — P-value is for Week 5; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 17: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.438, ANOVA — P-value is for Week 6; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 18: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.602, ANOVA — P-value is for Week 8; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 19: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.493, ANOVA — P-value is for Week 10; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 20: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.335, ANOVA — P-value is for Week 12; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 21: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.398, ANOVA — P-value is for Week 24; ANOVA with treatment, country, TZD use in the model
Statistical Analysis 22: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.903, ANOVA — P-value is for Endpoint; ANOVA with treatment, country, TZD use in the model

53. Secondary Outcome: ADDENDUM: Percentage of Participants With Self-reported Hypoglycemic Episodes
Description: Hypoglycemia = any time participant feels/person observes, that the participant is experiencing a sign/symptom they associate with hypoglycemia (such as hunger, dizziness, shakiness, light-headedness, sweating, irritability, headache, fast heart beat, confusion, etc) or a glucose measurement ≤70 mg/dL (≤3.9 mmol/L). Severe hypoglycemia = participant requires assistance. Qualified medical staff instructed the participants about the signs and symptoms of hypoglycemia.
Time Frame: Weeks 6 (Addendum: 30 weeks), 12 (36 weeks), 24 (48 weeks), Endpoint (LOCF)
Population: as for outcome 47
Measure: Number; unit: percentage of participants
Arm/Group | Basal Bolus Prior Lispro LM Addendum | Lispro Mid Mix Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum | Lispro Low Mix Prior Glargine Addendum
Number analyzed (Participants) | 164 | 171 | 192 | 198
percentage of participants
  Hypoglycemia episodes endpoint | 40.9 | 41.5 | 34.9 | 40.9
  Overall hypoglycemia episodes | 53.7 | 56.1 | 47.9 | 56.1
  Severe episodes endpoint | 0.0 | 0.0 | 0.0 | 0.0
  Severe episodes overall | 0.0 | 1.2 | 0.0 | 1.0
  Nocturnal episodes endpoint | 25.0 | 20.5 | 19.3 | 23.7
  Nocturnal episodes overall | 31.1 | 31.0 | 27.1 | 36.9
Statistical Analysis 1: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.953, Cochran-Mantel-Haenszel — P-value is for Hypoglycemia episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 2: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.953, Cochran-Mantel-Haenszel — P-value is for Overall hypoglycemia episodes; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 3: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.188, Cochran-Mantel-Haenszel — P-value is for Severe episodes overall; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 4: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.226, Cochran-Mantel-Haenszel — P-value is for Nocturnal episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 5: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.855, Cochran-Mantel-Haenszel — P-value is for Nocturnal episodes overall; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 6: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.250, Cochran-Mantel-Haenszel — P-value is for Hypoglycemia episodes at endpoint; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 7: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.123, Cochran-Mantel-Haenszel — P-value is for Overall hypoglycemia episodes; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 8: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.166, Cochran-Mantel-Haenszel — P-value is for Severe episodes overall; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 9: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.273, Cochran-Mantel-Haenszel — P-value is for Nocturnal episodes endpoint; Cochran-Mantel-Haenszel statistic controlling for country and TZD use
Statistical Analysis 10: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.039, Cochran-Mantel-Haenszel — P-value is for Nocturnal episodes overall; Cochran-Mantel-Haenszel statistic controlling for country and TZD use

54. Secondary Outcome: ADDENDUM: Rate of Self-reported Hypoglycemic Episodes
Description: Hypoglycemia = participant feels/person observes, that the participant is experiencing a sign/symptom they associate with hypoglycemia (such as hunger, dizziness, shakiness, light-headedness, sweating, irritability, headache, fast heart beat, confusion, etc) or a glucose measurement ≤70 mg/dL (≤3.9 mmol/L). Severe hypoglycemia = participant requires assistance. Qualified medical staff instructed the participants about the signs and symptoms of hypoglycemia.
Time Frame: Endpoint (Addendum 24 weeks), Overall (mean yearly rate of hypoglycemia during addendum phase
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: episodes/participant/year
Arm/Group | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro LM Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Number analyzed (Participants) | 171 | 198 | 164 | 192
episodes/participant/year
  Hypoglycemia episodes Endpoint | 11.10 (20.36) | 10.11 (21.84) | 12.11 (28.20) | 11.18 (44.80)
  Hypoglycemia episodes Overall | 11.54 (18.70) | 10.73 (18.06) | 11.39 (22.75) | 9.04 (21.45)
  Nocturnal episodes Endpoint | 2.46 (8.14) | 2.51 (7.03) | 2.37 (6.10) | 3.01 (13.62)
  Nocturnal episodes Overall | 2.47 (6.29) | 3.14 (6.58) | 2.09 (5.25) | 2.15 (5.56)
  Severe episodes Endpoint | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Severe episodes Overall | 0.02 (0.23) | 0.02 (0.21) | 0.00 (0.00) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.623, ANOVA — P-value is for Hypoglycemia episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 2: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.949, ANOVA — P-value is for Hypoglycemic episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 3: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.730, ANOVA — P-value is for Hypoglycemia episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 4: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.445, ANOVA — P-value is for Hypoglycemia episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 5: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.949, ANOVA — P-value is for Nocturnal episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 6: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.590, ANOVA — P-value is for Nocturnal episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 7: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.657, ANOVA — P-value is for Nocturnal episodes Endpoint; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 8: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.108, ANOVA — P-value is for Nocturnal episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 9: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.161, ANOVA — P-value is for Severe episodes Overall; Response = Treatment + Country + TZD use + Sulfo use
Statistical Analysis 10: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.178, ANOVA — P-value is for Severe episodes Overall; Response = Treatment + Country + TZD use + Sulfo use

55. Secondary Outcome: ADDENDUM: Change From Baseline in 1,5-Anhydroglucitol to Week 24
Time Frame: Baseline (addendum: 24 weeks), Endpoint (24 weeks: Week 48)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Basal Bolus Prior Lispro LM Addendum | Lispro Mid Mix Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum | Lispro Low Mix Prior Glargine Addendum
Number analyzed (Participants) | 166 | 172 | 197 | 199
ug/mL
  Baseline (n=166,172,197,199) | 7.84 (5.27) | 7.77 (5.01) | 7.31 (4.99) | 7.37 (5.07)
  Endpoint (n=142,150,165,171) | 8.18 (6.27) | 7.73 (5.74) | 8.43 (6.17) | 8.14 (5.21)
  Change (n=142,150,165,171) | 0.26 (4.40) | -0.18 (4.91) | 0.90 (4.31) | 0.53 (4.53)
Statistical Analysis 1: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.917, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 2: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.754, ANOVA — P-value for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 3: Comparison: Basal Bolus Prior Lispro LM Addendum vs Lispro Mid Mix Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.420, ANCOVA — P-value is for Change; ANCOVA model with treatment, baseline, country, and TZD use
Statistical Analysis 4: Comparison: Basal Bolus Prior Glargine Addendum vs Lispro Low Mix Prior Glargine Addendum; Test type: Superiority or Other; p = 0.514, ANCOVA — P-value for Change; ANCOVA model with treatment, baseline, country, and TZD use

56. Secondary Outcome: ADDENDUM: HbA1c at Specified Visits and Endpoint
Time Frame: Baseline (Addendum: 24 weeks), Weeks 12, 24, Endpoint (24 weeks: Week 48)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: percent glycosylated hemoglobin
Arm/Group | Lispro Mid Mix Prior Lispro Low Mix Addendum | Lispro LM Prior Glargine Addendum | Basal Bolus Prior Lispro Low Mix Addendum | Basal Bolus Prior Glargine Addendum
Number analyzed (Participants) | 174 | 200 | 171 | 199
percent glycosylated hemoglobin
  Baseline (n=174,200,171,199) | 8.01 (0.93) | 8.03 (0.95) | 8.00 (0.92) | 7.98 (0.95)
  Week 12 (n=150,175,151,161) | 8.11 (1.06) | 8.07 (1.20) | 8.13 (1.26) | 8.19 (1.38)
  Week 24 (n=145,171,144,159) | 8.19 (1.27) | 8.05 (1.18) | 8.19 (1.47) | 8.14 (1.55)
  Endpoint (n=160, 187,159,176) | 8.19 (1.26) | 8.03 (1.15) | 8.16 (1.43) | 8.14 (1.53)
Statistical Analysis 1: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.770, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 2: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.566, ANCOVA — P-value is for Week 12; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 3: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.812, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 4: Comparison: Lispro Mid Mix Prior Lispro Low Mix Addendum vs Basal Bolus Prior Lispro Low Mix Addendum; Test type: Superiority or Other; p = 0.990, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 5: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.552, ANOVA — P-value is for Baseline; ANOVA with treatment, country, TZD use in model
Statistical Analysis 6: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.179, ANCOVA — P-value is for Week 12; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 7: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.377, ANCOVA — P-value is for Week 24; Response = Treatment + Baseline + Country + TZD use
Statistical Analysis 8: Comparison: Lispro LM Prior Glargine Addendum vs Basal Bolus Prior Glargine Addendum; Test type: Superiority or Other; p = 0.271, ANCOVA — P-value is for Endpoint; Response = Treatment + Baseline + Country + TZD use

ADVERSE EVENTS:
Description: This trial did not collect non-serious adverse events other than hypoglycemia; results of which are included as secondary outcome measures.
Arm/Group | Insulin Glargine Initiation | Lispro LM Initiation | Lispro Mid Mix Prior Lispro LM Addendum | Lispro LM Prior Glargine Addendum | Basal Bolus Prior Lispro LM Addendum | Basal Bolus Prior Glargine Addendum | Insulin Glargine Maintenance | Lispro LM Maintenance
Serious Adverse Events (participants affected / at risk) | 45/1046 | 65/1045 | 5/174 | 10/200 | 9/171 | 11/199 | 48/419 | 48/473
Other Adverse Events (participants affected / at risk) | 785/1024 | 826/1026 | 96/171 | 111/198 | 88/164 | 92/192 | 394/419 | 463/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine Initiation (N=1046) | Lispro LM Initiation (N=1045) | Lispro Mid Mix Prior Lispro LM Addendum (N=174) | Lispro LM Prior Glargine Addendum (N=200) | Basal Bolus Prior Lispro LM Addendum (N=171) | Basal Bolus Prior Glargine Addendum (N=199) | Insulin Glargine Maintenance (N=419) | Lispro LM Maintenance (N=473)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Corneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail bed infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign female reproductive tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catatonia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine Initiation (N=1024) | Lispro LM Initiation (N=1026) | Lispro Mid Mix Prior Lispro LM Addendum (N=171) | Lispro LM Prior Glargine Addendum (N=198) | Basal Bolus Prior Lispro LM Addendum (N=164) | Basal Bolus Prior Glargine Addendum (N=192) | Insulin Glargine Maintenance (N=419) | Lispro LM Maintenance (N=473)
Hypoglycemia (Metabolism and nutrition disorders) | 785 (9994) | 826 (13164) | 96 (905) | 111 (927) | 88 (869) | 92 (785) | 394 (16861) | 463 (22562)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days